CLINICAL TRIAL: NCT05569655
Title: Efficacy and Safety Evaluation of Tolvaptan in the Treatment of Patients With Right Heart Failure Caused by Pulmonary Arterial Hypertension
Brief Title: Efficacy and Safety Evaluation of Tolvaptan in the Treatment of Patients With RHF Caused by PAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tolvaptan
Record Dates: First submitted 2022-10-01; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Arterial Hypertension; Randomized Controlled Trial
Keywords: Pulmonary arterial hypertension; Randomized controlled trial
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Tolvaptan; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects in group A (Experimental): For subjects in group A, tolvaptan (15 mg/d) is added to standard therapy (furosemide: 20mg-40mg/d).
  Interventions: Drug: Tolvaptan; Drug: Furosemide
- Subjects in group B (Active Comparator): Subjects in group B receive standard therapy (including furosemide: 20mg-40mg/d).
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Tolvaptan — Within 12 hours of admission, subjects were randomly assigned to two groups using the central randomization method. For subjects in group A, tolvaptan (15 mg/d) is added to standard therapy (furosemide:20-40mg/d). The treatment lasts for a total of seven days to assess the efficacy and safety of tolvaptan in the treatment of PAH-induced right heart failure.
  Other Names: Samsca
  Arms: Subjects in group A
Drug: Furosemide — Within 12 hours of admission, traditional standard therapy (furosemide:20-40mg/d) is used for all subjects in our clinical trial. The treatment lasts for a total of seven days.
  Other Names: LASⅨ

SUMMARY:
Efficacy and safety evaluation of tolvaptan in the treatment of patients with right heart failure caused by pulmonary arterial hypertension

DETAILED DESCRIPTION:
The study is a prospective, single-center, randomized controlled trial. Specifically, the research focuses on patients with right heart failure due to PAH in the Pulmonary Vascular Ward of Fuwai Hospital. Within 12 hours of admission, subjects were randomly assigned to two groups using the central randomization method. The dose of tolvaptan (15 mg/d) is added to standard therapy (including diuretics) for subjects in group A. Traditional standard therapy (including diuretics) is used for subjects in group B. The treatment lasts for a total of seven days to assess the efficacy and safety of tolvaptan in the treatment of PAH-induced right heart failure. An informed consent form must be signed by each participant in our study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have no serious cerebrovascular, liver, kidney and lung organ and tissue diseases.
* No corticosteroids or immunosuppressive agents had been administered to the - Patients in the three months prior to enrollment in the study.
* Patients voluntarily participated in the study and signed an informed consent form.

Exclusion Criteria:

* Patients who install the circulation aids.
* Patients who have been diagnosed with active myocarditis or amyloid cardiomyopathy.
* Fasting blood glucose level exceeded 12.21 mmol/L in individuals with uncontrolled diabetes.
* Patients who suffer from anuria, urethral strictures, stones, or tumors caused by urination disorders.
* Patients with acute myocardial infarctions, persistent ventricular tachycardias, or ventricular fibrillations, and cerebrovascular accidents within the first 30 days of the screening period.
* Patients with a history of allergy or specific reactions to benzodiazepines. (Mozavaputan hydrochloride, Benaepril hydrochloride)
* Any of the following laboratory tests were abnormal: serum creatinine> 2.5 times the upper normal value limit, serum sodium> 145 mmol/L, and serum potassium> 5.5 mmol/L.
* Pregnant women, lactating women, or patients who may be pregnant or have pregnancy plans.
* Patients with other contraindications to the use of tolvaptan.
* Patients who have been taking tolvaptan within the first 3 months before inclusion in the study, either when the drug was marketed or when it was being clinically studied.
* Additionally, patients who were judged by the investigators not fit to be enrolled in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight( in kilograms ) of 7 days after medication or discharge day(one earlier). | 7 days
  Changes in body weight ( in kilograms ) of 7 days after medication or discharge day(one earlier).
Changes in urine volume (in milliliters）of 7 days after medication or discharge day(one earlier). | 7 days
  Changes in urine volume ( in milliliters ) of 7 days after medication or discharge day(one earlier).

SECONDARY OUTCOMES:
Blood creatinine changes in renal function. | 7 days
  Blood creatinine changes in renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD#PhD, Study Director — center of pulmonary vascular disease, Fuwai hospital
Locations (1):
- center of pulmonary vascular disease, Fuwai hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No